CLINICAL TRIAL: NCT06783036
Title: Long-term Recurrence and Other Complications Requiring Surgery Following Primary Ventral Hernia Repair
Status: Active, not recruiting | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Erling Oma, Principal Investigator, Bispebjerg Hospital
Other Study IDs: P-2023-193; R-23045342 (Other: Team for journaldata, Center for sundhed); DHDB-2023-04-03 (Other: Dansk herniedatabase); FSEID-00006723 (Other: Sundhedsdatastyrelsen)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Umbilical Hernia; Epigastric Hernia
MeSH Terms: conditions — Hernia, Umbilical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Emergency umbilical hernia repair: no study intervention
- Elective umbilical hernia repair: no study intervention
- Emergency epigastric hernia repair: no study intervention
- Elective epigastric hernia repair: no study intervention

SUMMARY:
Nationwide, registry based cohort studies on all complications requiring surgery following primary ventral hernia repair

DETAILED DESCRIPTION:
Cohort based on patients registered in the Danish Ventral Hernia Database. Through cross-linking at an individual level, all subsequent operations will be identified in the Danish National Patient Registry. For all potentially related reoperations, patient charts will be retrieved and manually reviewed. Furthermore cross-linkage with the Danish Civil Registration System to retrieve information on civil status. Follow up from time of operation for primary ventral hernia repair (index operation) until reoperation, death, emigration or end of follow up (December 31, 2023), whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Operation for primary ventral hernia repair registered in Danish Ventral Hernia Database
* Known body mass index and smoking status at time of surgery, as registered in the Danish Ventral Hernia Database

Exclusion Criteria:

* Hernia type misclassification (based on manual medical file review)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nationwide population of patients registered in the Danish Ventral Hernia Database
Sampling Method: Non-Probability Sample
Enrollment: 7200 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Operation for hernia recurrence | Until december 31, 2023

SECONDARY OUTCOMES:
Operation for non-recurrence complication | Until december 31, 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Digestive Disease Center, Bispebjerg Hospital, Copenhagen, Denmark